CLINICAL TRIAL: NCT06299722
Title: Strength Training Exercises to Minimise Late Effects of Childhood Leukaemia or Lymphoma Among Adolescents - The STEEL Study - a National Multicenter Randomised Controlled Study
Brief Title: Strength Training Exercises to Minimise Late Effects of Childhood Leukaemia or Lymphoma Among Adolescents
Acronym: STEEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Riel, Postdoctoral researcher, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20230055
Record Dates: First submitted 2024-02-14; First posted 2024-03-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Steel; Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEEL (Experimental): STEEL strength training will consist of progressive periodised training, in which the intensity is set to fit the individual's starting level and then gradually increases. During Week 1 to Week 5, the relative load will correspond to a 12-repetition maximum (RM). During Week 5 to Week 10, the relative load will be 10 RM, and during Week 11 to Week 16, the relative load will be 8 RM. The exercises will mostly consist of compound movements that activate the large muscle groups of the legs, back, arms and torso.
  Interventions: Other: STEEL
- Circuit training (Active Comparator): There will be 10 stations that include both strengthening and cardiovascular exercises, such as squats, hopping, crunches, stationary running, front-lying swimming, ski jumps, push-ups, ball throws, ring pulls, and hopscotch. Each station lasts 45 seconds, and there will be a 15-second break between each station. The circuit is repeated for three rounds. To ensure progression in intensity similar, we will progress the participants' rating of perceived exertion (RPE) over time. During Week 1 to Week 5, the RPE during exercises will be 6-7. During Week 5 to Week 10, the RPE will be 8-9, and during Week 11 to Week 16, the RPE will be 10.
  Interventions: Other: Circuit training

INTERVENTIONS:
Other: STEEL — Relatively heavy strength training
  Arms: STEEL
Other: Circuit training — Circuit training
  Arms: Circuit training

SUMMARY:
We aim to include 60 children and adolescents aged 10 to 19 years who have undergone successful treatment for leukemia or lymphoma. Based on randomization, they will either 1) commence 16 weeks of training with STEEL or 2) commence 16 weeks of circuit training. STEEL training involves exercises for major muscle groups using free weights, body weight, or tailored machines. Circuit training is structured similarly to previous training for the target group and includes exercises using body weight, exercise balls, and rings. The training takes place in local centers either with friends or with other participants in the project. Before starting participation in the project, the child/adolescent and their parents or guardians will receive information about late effects, diet, sleep, and exercise, providing guidance and support regarding the project elements. The effects of the two training modalities will be evaluated based on self-reported quality of life, muscle strength, muscle mass, bone mineral content, fitness, and markers of metabolic syndrome (BMI, waist circumference, blood pressure, and blood analysis).

DETAILED DESCRIPTION:
The trial is designed as a national randomised clinical trial. Participants will be stratified by sex and block randomised (block sizes of 2 to 6) at 1:1 to either STEEL or the circuit training programme. A researcher not involved in the trial will generate the allocation sequence using a random number generator and is the only person who will know the block sizes. The study will be conducted at Aalborg University Hospital, Rigshospitalet, Odense University Hospital, and Aarhus University Hospital and was designed in collaboration with parents of childhood cancer survivors and an adult childhood cancer survivor suffering from late effects. Participants must attend three examinations at their respective hospitals: baseline and after 8 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ten to 19 years of age at the point of inclusion
* A minimum of 12 months since the last chemotherapy with no upper limit
* Ability to understand the physical intervention and general participant advice

Exclusion Criteria:

* Participation in another research study that includes similar treatment
* Pregnancy
* Cardiac arrhythmia during exercise
* Psychological disorders interfering with treatment
* Presence of a clinical condition that needs immediate treatment
* Planned surgeries within the subsequent 12 months that may interfere with performing exercises
* Any contraindications to performing physical exercise as evaluated by the recruiting medical doctor

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Isometric strength | Baseline and at the 8-week and 16-week follow-ups
  Measured in Nm based on tests of knee extension and flexion and elbow extension and flexion using handheld dynamometry

SECONDARY OUTCOMES:
Health-related quality of life | During baseline and at the 16-week follow-up
  We will use the Danish version of the Pediatric Quality of Life Inventory (PedsQL™) 4.0 Generic Core scales and the PedsQL™ Multidimensional Fatigue scales (5,9) to assess health-related quality of life. The PedsQL is a brief 23-item measurement model that evaluates quality of life in four areas: physical, emotional, social and school functioning. The questionnaire scores range from 0 to 100, and higher scores indicate better quality of life. The PedsQL™ Multidimensional Fatigue includes 18 questions related to fatigue and uses the same scoring as the PedsQL
Step counts | Weekly throughout the 16-week intervention
  We will assess participants' step counts throughout the intervention using a Garmin vívosmart® 5 watch (Garmin Ltd., Kansas, USA).
Caloric expenditure | Weekly throughout the 16-week intervention
  We will assess participants' caloric expenditure (KCAL) throughout the intervention using a Garmin vívosmart® 5 watch (Garmin Ltd., Kansas, USA).
Maximal dynamic strength | During the first and last training sessions of the 16-week intervention
  we will test the 1 repetition maximum (RM) in the leg press and chest press machines
Bone mineral density of the lumbar spine and body composition | During baseline and at the 16-week follow-up
  We will measure the bone mineral density of the lumbar spine (L1-L4) calculated as the Z-score and body composition (%body fat, lean body mass, and skeletal muscle mass) by a dual-energy-X-ray absorptiometry scanner located at each hospital.
Grip strength and rate of force development | Baseline and at the 8-week and 16-week follow-ups
  Using a digital hand dynamometer, we will measure continuous isometric handgrip force and rate of force development.
Muscular strength, endurance, and rate of force development | Baseline and at the 8-week and 16-week follow-ups
  We will use a 30-second sit-to-stand test to evaluate strength, endurance, and rate of force development of the lower extremities.
Cardiorespiratory fitness and endurance | Baseline and at the 8-week and 16-week follow-ups
  We will perform a 6-minute walk test to evaluate cardiorespiratory fitness and walking endurance
Exercise compliance and fidelity | Throughout the 16-week intervention
  Exercise compliance and fidelity will be measured using training diaries, which the participants fill out themselves after the unsupervised training sessions and by the physiotherapist during the supervised training sessions. Exercise compliance relates to whether the training sessions have been performed, and fidelity relates to whether the exercises have been performed as prescribed regarding the number of repetitions, sets, and intensity.
Adverse events | Throughout the 16-week intervention
  Adverse events will be collected throughout the trial and graded 1 to 5 according to the Common Terminology Criteria for Adverse Events v4.03. Participants are asked to contact the responsible clinician at the hospital where they were enrolled as soon as they experience any adverse event.
Movement-evoked pain | During baseline and at the 16-week follow-up
  We will use a 0 (no pain) to 10 (worst pain imaginable) Numerical Rating Scale to assess movement-evoked pain during the past week
Satisfaction with the intervention | During the 16-week follow-up
  We will assess participant satisfaction with their respective intervention using a 5-point rank scale ranging from 'very dissatisfied' to 'very satisfied'.
Blood glucose | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/L
Glycated hemoglobin (Hba1c) | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/mol
Insulin | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mU/L
Proinsulin c-peptide | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in ng/mL
Total cholesterol | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/L
High-density lipoprotein cholesterol | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/L
Low-density lipoprotein cholesterol | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/L
Very low-density lipoprotein cholesterol | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/L
Triglycerides | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in mmol/L
Glucagon | During baseline and at the 16-week follow-up
  Analysed from a blood sample and measured in pg/mL
Homeostatic Model assessment for Insulin resistance score | During baseline and at the 16-week follow-up
  Calculated as fasting plasma glucose (mmol/L x fasting plasma glucose ((μU/L)/22.5) to estimate β-cell function (HOMA-B) and insulin-resistance (HOMA-IR2)
Body Mass Index (BMI) | During baseline and at the 16-week follow-up
  Measured as kg/m² for adolescents aged 18 or 19 years and BMI standard deviation (SD) scores for children aged 10-17 years based on national reference material.
Lean body mass | During baseline and at the 16-week follow-up
  Measured in kilograms based on dual-energy X-ray absorptiometry (DXA)
Fat mass | During baseline and at the 16-week follow-up
  Measured in kilograms based on dual-energy X-ray absorptiometry (DXA)
Android/gynoid fat distribution | During baseline and at the 16-week follow-up
  Measured in kilograms based on dual-energy X-ray absorptiometry (DXA) adjusted for sex and pubertal stage
Abdominal circumference | During baseline and at the 16-week follow-up
  Measured in centimetres
Self-reported Tanner staging | During baseline and at the 16-week follow-up
  Visual illustration of Tanner staging (I-V) regarding both genders
Blood pressure | During baseline and at the 16-week follow-up
  Measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Madeleine, DSc, Study Chair — Aalborg University
Locations (4):
- Denmark (4):
  - Århus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Aalborg University, Gistrup
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP